CLINICAL TRIAL: NCT00940979
Title: Prospective Randomised Trial Using Integuseal as Microbial Sealant for Arterial Bypass Surgery on Lower Extremities
Brief Title: Trial Using Integuseal as Microbial Sealant for Arterial Bypass Surgery on Lower Extremities
Acronym: ITT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analyses showed insufficient result. Termination for reasons of futility
Sponsor: Rijnstate Hospital (Other)
Collaborators: Kimberly-Clark Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LTC 625-230609
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Arterial Obstructive Diseases
Keywords: Integuseal microbial sealant; Infection prophylaxis; Postoperative wound infection; Arterial bypass surgery
MeSH Terms: conditions — Arterial Occlusive Diseases; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- No use of integuseal (No Intervention)
- Use of Integuseal (Experimental): Application of a layer of Integuseal (Cyanoacrylate) from a ready to use applicator preoperative before incision Polymerisation immobilise the bacteria that survived the conventional skin preparation This way there will be les contamination of the wound.
  Interventions: Procedure: Application of Integuseal sealant

INTERVENTIONS:
Procedure: Application of Integuseal sealant — Microbial sealant (integuseal) applied with a sponge applicator
  Arms: Use of Integuseal

SUMMARY:
The purpose of this study is to prove a reduction of postoperative wound infections after direct preoperative use of a microbial sealant in the form of Integuseal for vascular procedures on lower extremities.

ELIGIBILITY:
Inclusion Criteria:

* planned supragenual of infragenual peripheral arterial bypass procedures with autologue or prosthetic graft

Exclusion Criteria:

* secondary procedures and suprainguinal procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Postoperative wound infections

SECONDARY OUTCOMES:
Costs of the use of Integuseal
Complications during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Michel MPJ Reijnen, MD, Study Director — Rijstate hospital Arnhem the Netherlands; J. Klinkenbijl, MD, Study Director; Sjoerd A de Beer, MD, Principal Investigator — Rijnstate Hospital Arnhem the Netherlands
Locations (3):
- Netherlands (3):
  - Ziekenhuis Rijnstate, Arnhem
  - Ziekenhuis Slingland, Doetinchem
  - Ziekenhuis Nij Smellinghe, Drachten